CLINICAL TRIAL: NCT05640063
Title: Evaluation of the Impact of Enhanced Delivery and Newborn Kits as Compared to Standard Delivery Kits in the Flood Affected Districts of Sindh and Balochistan Provinces: A Cluster Randomized Trial
Brief Title: Evaluation of Enhanced Delivery and Newborn Kit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Distinguish University Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0979-3131
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Perinatal Death
Keywords: perinatal mortality; delivery kit; Newborn kit; health services
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Intervention Model Description: We are considering Union Council as a cluster. Clusters will be identified and matched on population size, socio-economic status (including structure, electricity, drinking water assets with HH density), birth/death rates, and number of functional LHWs and CMWs. Paired randomization will be done to allocate one group (intervention/control) to each cluster and all the LHWs in one union council will be assigned to one group to avoid any sort of contamination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Provision of Enhanced Delivery and Newborn Kits (CMWs and LHW program will continue to function as usual)
  Interventions: Other: Enhanced Delivery and Newborn kit
- Control Arm (No Intervention): Standard Delivery Kits alone (CMWs and LHW program will continue to function as usual)

INTERVENTIONS:
Other: Enhanced Delivery and Newborn kit — Under this study enhanced delivery and newborn kits will be provided to the identified pregnant women to utilize at home or at health facility and avoid delays at facility. After the training of community and health care providers, the intervention package will be delivered in the intervention clusters primarily through the LHWs and CMWs.
  Arms: Intervention Arm

SUMMARY:
The evidence is required to assess the effectiveness of enhanced delivery and newborn kits as compared to standard delivery kits in the flood affected districts that can increase the utilization of services and reduce the delays that are responsible for poor maternal and newborn health through LHW program.

DETAILED DESCRIPTION:
Addressing birth-related deaths is especially important since they frequently result from problems during childbirth, creating emergency situations with a limited window of opportunity for intervention (1).Globally, 2.4 million newborns die each year with one million of these neonatal deaths in the first week of life and 1.2 million stillborn neonates are caused by maternal health complications, indicating a significant intervention gap exists throughout pregnancy, childbirth, and the early postpartum period, when mothers and babies are most at risk (2). The major cause of maternal mortality is obstetric hemorrhage, puerperal sepsis, and hypertensive disorders in pregnancy. Anemia and malaria are the commonest indirect cause of maternal morbidity and mortality (3). Among newborn deaths sepsis is the leading cause followed by birth asphyxia and low birth weight. These complications compounded by unhygienic delivery practices such as lack of cord care, with no proper handwashing and improper waste disposal at home and at facility (4).

Though, there are many variables that contribute to maternal and neonatal fatalities, one of the most efficient ways to address this issue is to quickly provide mothers and newborns with effective preventive measures or treatment, frequently at home or at first level healthcare platform (5; 6).

Recent rains and floods also have damaged not only the health care facilities but access to these facilities is a challenge (10). In times of crisis, the capacity of health facilities, including skilled birth attendants and emergency obstetric care is often unavailable, which increases women's vulnerability. Complications that occur during pregnancy or childbirth are a leading cause of death and illness among women and young girls in the affected areas. According to the United Nations Population Fund, more than 650,000 pregnant women in flood affected areas require urgent maternal health services, with at least 73,000 women expected to give birth. (11).Hypothesis We hypothesize that provision of the Enhanced delivery and newborn kits will reduce the Perinatal mortality as compared to standard delivery kits Operational Definition of Perinatal Mortality "Perinatal mortality is an important outcome indicator for newborn care and directly mirrors the quality of prenatal, intra partum and newborn care" (18).

The specific objectives of this study are

Primary Objective:

• To reduce the perinatal mortality in flood affected areas

Secondary Objectives:

* To mobilize community for creation of demand for improved MNH services and practices through community mobilization.
* To increase knowledge of target audiences for pregnancy, delivery, postdelivery and newborn danger signs
* To increase clean deliveries at home through provision of enhanced delivery and newborn kits
* To improve newborn care practices
* To strengthen and improve the quality of maternal and newborn care at health facilities through referral linkages Methodology Study design Cluster randomized controlled trial. Study Site and Context The Study will be conducted in in the flood affected districts (Lasbella, Qamabr Shahdad Kot, Sanghar and Dadu) within the Umeed e Nau (UeN) project Balochistan & Sindh. The project is operational in these areas through field offices. Maternal, Newborn and Child Health (MNCH) focused interventions are already rolled out, including capacity building of health care providers at secondary level care public health facility and community level on MNCH services i.e., EmONC, IMNCI (Integrated Management of Newborn and Child illness) and IYCF (Infant and young child feeding). The project field teams include doctors, social mobilizers, and technical personnel for the implementation of activities in close liaison with department of health (DOH).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the project sites living in the area till expected date of their delivery.

Exclusion Criteria:

* The individuals who would not consent to participate in the study voluntarily.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Perinatal mortality rate | 12 months
  "Perinatal mortality is an important outcome indicator for newborn care and directly mirrors the quality of prenatal, intra partum and newborn care"

SECONDARY OUTCOMES:
Cause specific neonatal mortality | 12 months
  such as deaths related to omphalitis, birth asphyxia, prematurity, and sepsis.
Cause specific maternal mortality | 12 months
  such as deaths related to postpartum hemorrhage, puerperal sepsis, eclampsia, obstructed labor, unsafe abortion, and indirect causes (anemia, malaria)
Maternal morbidity | 12 months
  such as (including obstetric fistula, eclampsia, and obstetrical sepsis)

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No